CLINICAL TRIAL: NCT07022249
Title: Efficacy and Safety of a Novel Intrasaccular Embolization Device for the Treatment of Intracranial Aneurysms : a Prospective, Multicenter, Single-arm Trial
Brief Title: Evaluation of a Novel Intrasaccular Embolization Device for the Treatment of Intracranial Aneurysms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ202501
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Intrasaccular Embolization Device
  Interventions: Device: Intrasaccular Embolization Device

INTERVENTIONS:
Device: Intrasaccular Embolization Device — This is an intra-aneurysmal device intended for use in endovascular embolization of intracranial aneurysms.The intended therapeutic effect of this device is to line the neck of the aneurysm with a metallic structure that disrupts the inflow of blood, causing hemostasis within the aneurysm sac, and leading to thrombus formation within the implant.

SUMMARY:
The study is a prospective, multicenter single-arm cohort. The purpose of this study is to evaluate efficacy and safety of a novel intrasaccular embolization device for the treatment of intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18-75 years of age at the time of screening.
* Patient must have a single ruptured or unruptured IA requiring treatment.
* Patient was able to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule, signed and dated an written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Patient had an IA with characteristics unsuitable for endovascular treatment.
* Patient had vessel characteristics, tortuosity or morphology which precluded safe access and support during treatment with study device.
* Patient had vascular disease or other vascular anomaly that precluded the necessary access to the aneurysm for use of the study device.
* Patient had vasculitis, an intracranial tumor (except benign tumors that do not require treatment) or any other intracranial vascular malformations on presentation.
* Patient was taking anticoagulants or had a known blood dyscrasia, coagulopathy, or hemoglobinopathy.
* Patient was pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The Primary Safety Endpoint Included Any Death or Major Stroke in the First 30 Days and Neurologic Death or Ipsilateral Major Stroke Between Day 31 and Day 365. | 12 months
Percentage of Subjects With Complete Aneurysm Occlusion Without Retreatment, Recurrent Subarachnoid Hemorrhage, Without Significant Parent Artery Stenosis (>50% Stenosis) at One Year After Treatment. | 12 months

IPD SHARING:
Plan to Share IPD: Undecided